CLINICAL TRIAL: NCT01596686
Title: Comparison of Preparation Regimens for Colonoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinical Hospital Colentina (Other)
Responsible Party: Principal Investigator, dr. Theodor Alexandru Voiosu, gastroenterology resident, Clinical Hospital Colentina
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: COL-GASTRO-2
Record Dates: First submitted 2012-05-07; First posted 2012-05-11 (Estimated); Last update posted 2013-12-24 (Estimated); Status verified 2013-12

CONDITIONS: Colonoscopy Preparation
MeSH Terms: interventions — picosulfate sodium

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- sodium picosulphate and magnesium citrate (Picoprep) (Active Comparator)
  Interventions: Drug: one of two possible colon preparation regimens
- polyethylene glycol (Fortrans) (Active Comparator)
  Interventions: Drug: one of two possible colon preparation regimens

INTERVENTIONS:
Drug: one of two possible colon preparation regimens — Patients are randomized to receive one of the two different preparation regimens for colonoscopy usually employed in our unit, polyethylene glycol or sodium picosulphate and magnesium citrate
  Other Names: Fortrans; Picoprep

SUMMARY:
The investigators intend to study the impact of two different preparation regimens for colonoscopy (PEG vs sodium picosulphate) on the quality of the endoscopy as well as patient tolerability.

ELIGIBILITY:
Inclusion Criteria:

* all patients undergoing colonoscopy

Exclusion Criteria:

* patient refusal to sign informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Actual)
Dates: Start 2012-05; Primary Completion 2012-12 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
colon preparation | 24 h
  the impact of colon preparation as assessed by the endoscopist (scale from 1 to 4, 1 representing the worst and 4 the best prepared colon) on the quality of the endoscopic examination

CONTACTS AND LOCATIONS:
Locations (2):
- Romania (2):
  - Colentina Clinical Hospital, Bucharest, Bucharest
  - Spitalul clinic judetean, Timișoara, Timisoara

REFERENCES:
- [Background] Manno M, Pigo F, Manta R, Barbera C, Bertani H, Mirante VG, Dabizzi E, Caruso A, Olivetti G, Hassan C, Zullo A, Conigliaro R. Bowel preparation with polyethylene glycol electrolyte solution: optimizing the splitting regimen. Dig Liver Dis. 2012 Jul;44(7):576-9. doi: 10.1016/j.dld.2012.02.012. Epub 2012 Mar 26. PMID 22456624
- [Result] Voiosu T, Ratiu I, Voiosu A, Iordache T, Schipor A, Baicus C, Sporea I, Voiosu R. Time for individualized colonoscopy bowel-prep regimens? A randomized controlled trial comparing sodium picosulphate and magnesium citrate versus 4-liter split-dose polyethylene glycol. J Gastrointestin Liver Dis. 2013 Jun;22(2):129-34. PMID 23799210